CLINICAL TRIAL: NCT05134441
Title: A Multi-Center, Randomized, Double-Blinded Phase 3 Study to Evaluate the Efficacy, Safety, and Tolerability of IMU-838 Versus Placebo in Adults With Relapsing Multiple Sclerosis (ENSURE-1)
Brief Title: Study to Evaluate the Efficacy, Safety, and Tolerability of IMU-838 in Patients With Relapsing Multiple Sclerosis
Acronym: ENSURE-1
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Immunic AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P3-IMU-838-RMS-01
Record Dates: First submitted 2021-09-30; First posted 2021-11-26 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- IMU-838 (Experimental): IMU-838 (vidofludimus calcium), a small molecule inhibitor of DHODH.
  Formulation:
  Tablets with 15 or 30 mg IMU-838 for once daily oral intake in the morning.
  Interventions: Drug: IMU-838 tablets
- Placebo (Placebo Comparator): Matching placebo, as described for the test product, identical number of tablets as given for IMU-838.
  Interventions: Drug: Placebo matching IMU-838 tablets

INTERVENTIONS:
Drug: IMU-838 tablets — Patients are randomized to IMU-838 or placebo in ratio 1:1
  Other Names: vidofludimus calcium
  Arms: IMU-838
Drug: Placebo matching IMU-838 tablets — Patients are randomized to IMU-838 or placebo in ratio 1:1
  Other Names: Placebo matching vidofludimus calcium
  Arms: Placebo

SUMMARY:
Multi-Center, Randomized, Double-Blinded Phase 3 Study to Evaluate the Efficacy, Safety, and Tolerability of IMU-838 versus Placebo in Adults with Relapsing Multiple Sclerosis (ENSURE-1)

DETAILED DESCRIPTION:
This study will be a multicenter, randomized, double-blind, placebo-controlled study with a blinded Main Treatment Period (MT) and an Open Label Period (OLE) to evaluate the efficacy, safety, and tolerability of IMU-838 in adult patients with RMS. The study will consist of the following periods:

Screening Period: Approximately 28 days Main Treatment Period: Up to 72 weeks (approximately 15 months) Open Label Extension Period: Up to approximately 8 years

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient (age ≥18 to ≤55 years).
* Patients with an established diagnosis of MS according to 2017 McDonald Criteria.
* Patients with RMS comprising of relapsing remitting MS (RRMS) and active secondary progressive MS, both defined according to Lublin criteria 1996 and 2014.
* Active disease as defined by Lublin 2014 evidenced prior to Screening by:

  1. At least 2 relapses in the last 24 months before randomization, or
  2. At least 1 relapse in the last 12 months before randomization, or
  3. A positive Gd+ MRI scan (brain and/or spine) in the last 12 months prior to randomization.
* Willingness and ability to comply with the protocol.
* Written informed consent given prior to any study-related procedure.

Exclusion Criteria:

* Patients with non-active secondary progressive MS and primary progressive MS.
* Any disease other than MS that may better explain the signs and symptoms, including history of complete transverse myelitis.
* Clinical signs or presence of laboratory findings suggestive for neuromyelitis optica (NMO) spectrum disorders or myelin oligodendrocyte glycoprotein (MOG)-IgG-associated encephalomyelitis
* Any active and uncontrolled coexisting autoimmune disease, other than MS (except for type 1 diabetes mellitus and inflammatory bowel disease)
* Use of experimental/investigational drug (with the exception ofCOVID-19 vaccines approved by emergency use authorization) and/or participation in drug clinical studies within 6 months prior to Screening
* Previous or current use of MS treatments lifelong, or within a pre-specified time period.
* Use of the pre-specified concomitant medications.
* Clinically significantly abnormal and pre-specified lab values.
* History of chronic systemic infections within 6 months before the date of informed consent.
* Diagnosis or suspected liver function impairment, which may cause fluctuating liver function tests during this study.
* Known history of nephrolithiasis or underlying condition with a strong association of nephrolithiasis.
* History or clinical diagnosis of gout.
* History or presence of any major medical or psychiatric illness
* Substantial medical condition that could create undue risk to the patient, could affect adherence with the study protocol or could undesirably affect study outcomes

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1050 (Estimated)
Dates: Start 2021-11-18 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2032-09 (Estimated)

PRIMARY OUTCOMES:
To evaluate efficacy of IMU-838 versus placebo regarding time to first relapse | 72 weeks
  Survival analysis of time to first relapse, occurred after the start of study treatment administration and before the end of the double-blind period, censored at a maximum of 72 weeks.

SECONDARY OUTCOMES:
Effect of IMU-838 versus placebo on volume of new T2 lesions | 72 weeks
  To evaluate the effect of IMU-838 versus placebo on volume of new T2 lesions. Mean difference between IMU-838- and placebo in changes of the volume of new MRI T2 lesions over 24-weeks of treatment in the double-blind period.
Effect of IMU-838 versus placebo on disability progression | 72 weeks
  To evaluate the effect of IMU-838 versus placebo on disability progression. Survival analysis of time to 12-week confirmed disability progression, as measured on Expanded Disability Status Scale during the double-blind period, censored at maximum 72-weeks.
Effect of IMU-838 versus placebo on cognitive performance | 72 weeks
  To evaluate the effect of IMU-838 versus placebo on cognitive performance. Survival analysis of time to confirmed clinically relevant changes on Symbol Digit Modalities Test during the double-blind period, censored at maximum 72-weeks.
Effect of IMU-838 versus placebo on whole brain atrophy | 72 weeks
  To evaluate the effect of IMU-838 versus placebo on whole brain atrophy. Difference in the mean of the percentage change on the whole brain volume between IMU-838 and placebo during the 72-weeks double-blind period.
Safety of IMU-838 versus placebo | 72 weeks
  To evaluate safety and tolerability of IMU-838 versus placebo by assessing rates of Treatment Emergent Adverse Events, Adverse Events of Special Interest, Serious Adverse Events, changes in levels of pre-specified laboratory parameters, vital signs and ECG parameters and rates and reasons for study discontinuations.

CONTACTS AND LOCATIONS:
Overall Officials: Robert J. Fox, MD, Principal Investigator — Mellen Center for MS, Neurological Institute, Cleveland Clinic, Ohio
Locations (86):
- United States (6):
  - Xenoscience, Inc., 21st Century Neurology, Phoenix, Arizona
  - Bradenton Research Center, Bradenton, Florida
  - Reliant Medical Research, LLC, Miami, Florida
  - Collier Neurologic Specialists, Naples, Florida
  - Neurology Associates of Ormond Beach, Ormond Beach, Florida
  - Consultants in Neurology, Ltd, Northbrook, Illinois
- Albania (2):
  - Klinika Mjekesore Nuova, Neurology Clinic, Tirana
  - Hygeia Hospital Tirana, Tirana
- Bulgaria (22):
  - MHAT Puls AD, Blagoevgrad
  - MHAT "Heart and Brain", EAD, Burgas
  - MC Exacta Medica OOD, Pleven
  - MHAT Avis Medica, Pleven
  - UMHAT Dr.Georgi Stranski EAD, Pleven
  - Heart and Brain University Hospital, Pleven
  - MC Vita 1, Pleven
  - UMHAT Sveti Georgi, Plovdiv
  - UMHAT "Medica Ruse", Rousse
  - CCB Medical Institute Ministry of Interior, Sofia
  - Diagnostic and Consultative Center Neoclinic, Sofia
  - UMHAT "Sveti Ivan Rilski" EAD, Sofia
  - MHATNP "Sveti Naum", EAD, Sofia
  - MHATNPsy Sveti Naum EAD, Sofia
  - UMHAT "Alexandrovska" EAD, Sofia
  - UMHAT "Alexandrovska", Sofia
  - Military Medical Academy MHAT, Sofia
  - MHAT "Sveta Sofia" EOOD, Sofia
  - Military Medical Academy, Sofia
  - UMHAT"Tsaritsa Yoanna -ISUL, Sofia
  - UMHATEM N.Pirogov, Sofia
  - UMHAT "Sveta Marina" EAD, First Clinic of Neurological Diseases, Varna
- Colombia (2):
  - Clínica Colsanitas S.A. Sede Clínica Universitaria Colombia, Bogotá
  - Neurocountry Portoazul S.A.S., Puerto Colombia
- Georgia (10):
  - 1st Uni Clinic of Tbilisi LEPL, Tbilisi
  - Eristavi Experimental Center, Tbilisi
  - J.S.C. Curatio Clinic, Tbilisi
  - Katsiashvili Emergency Center, Tbilisi
  - Khechinashvili University Hospital, Tbilisi
  - LTD Aversi Clinic, Tbilisi
  - LTD New Hospitals, Tbilisi
  - MediClub Georgia LLC, Tbilisi
  - Pineo Medical Ecosystem LTD, Tbilisi
  - Sarajishvili Neurology Institute, Tbilisi
- Greece (2):
  - Athens Medical Center, Athens
  - Thessaloniki Hosptl, Thessaloniki
- India (7):
  - Kanoria Hospital & Research Centre, Gandhinagar
  - Mallikatte, Kadri, Mangalore
  - Jasleen Hospital, Nagpur
  - Sir Ganga Ram Hospital, New Delhi
  - Ruby Hospital, Pune
  - Indira Gandhi Medical College & Hospital, Shimla
  - Institute of Medical Sciences Banaras Hindu University,IMS BHU Varanasi, Varanasi
- Jordan (2):
  - TSH Advanced Clinical Center, Amman
  - Irbid Speciality Hospital, Irbid
- Lebanon (2):
  - Hotel Dieu de France Hospital, Beirut
  - AUB Medical Center, Hamra
- Lithuania (2):
  - Lietuvos Sveikatos Mokslu Universitetas - Kauno Klinikos, Kaunas
  - Klaipedos Universitetine Ligonine - Klaipedos Issetines Sklerozes Centra, Klaipėda
- Mexico (9):
  - Neurociencias Estudios Clínicos S.C, Culiacán
  - Instituto Jalisciense de Metabolismo, SC, Guadalajara
  - Grupo medico camino SC, Mexico City
  - Cliditer S.A de C.V, Mexico City
  - Unidad de Investigación en Salud de Chihuahua S.C., Mexico City
  - Clinstile SA de CV, Mexico City
  - Centro de Morelia, Morelia
  - Faicic de RL de CV, Veracruz
  - Sociedad de Metabolismo y Corazon, S.C., Veracruz
- Moldova (3):
  - Instititute of Emergency Medicine, Chisinau
  - Medico-Sanitary Public Institution, Institute of Neurology and Neurosurgery "Diomid Gherman", Chisinau
  - The Diomid Gherman Institute of Neurology and Neurosurgery, Chisinau
- Montenegro (2):
  - General Hospital Niksic, Nikšić
  - Clinical Center of Montenegro, Podgorica
- North Macedonia (2):
  - Hospital "8 mi Septemvri", Skopje
  - University Clinic of Neurology, Skopje
- Hospital Universitario La Paz, Madrid, Spain
- Ukraine (12):
  - Chernihiv Regional Hospital, Chernivtsi
  - Regional Clinical Hospital, Ivano-Frankivsk
  - Neuro Global, LLC, Ivano-Frankivsk
  - Khmelnytsky regional hospital of war veterans, Khmelnytskyi
  - Clinical Hospital #15 of the Podilskyi District of the Kyiv City, Kiev
  - "Medbud", Kyiv
  - SMART medical center, Kyiv
  - Kyiv City Hospital 4, Kyiv
  - Odesa Regional Clinical Hospital, Department of Neurosurgery, Odesa
  - Medical and diagnostic center of a LLC "Medcontinent", neurology and rehabilitation center, Poltava
  - Ternopil Psycho-Neuro Hospital, Ternopil
  - Regional Clinical Center for Neurosurgery and Neurology, Uzhhorod

IPD SHARING:
Plan to Share IPD: No